CLINICAL TRIAL: NCT00351884
Title: A Multicenter, Double-blind, Randomized, Parallel-Group Study to Compare the Effect of 24 Weeks Treatment With Vildagliptin 100 MG QD to Placebo as Add-on Therapy in Patients With Type 2 Diabetes Inadequately Controlled With Metformin Monotherapy
Brief Title: Efficacy of Vildagliptin 100 MG as Compared to Placebo as Add-on to Metformin in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals Corporation
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLAF237A23103
Record Dates: First submitted 2006-07-11; First posted 2006-07-13 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes; vildagliptin; Hemoglobin A1c
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- vildagliptin am (Experimental)
  Interventions: Drug: Vildagliptin AM
- vildagliptin pm (Experimental)
  Interventions: Drug: vildagliptin pm
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Vildagliptin AM
  Arms: vildagliptin am
Drug: vildagliptin pm
  Arms: vildagliptin pm
Drug: placebo
  Arms: placebo

SUMMARY:
Vildagliptin is an oral anti-diabetic agent. This is a 24-week study to assess the efficacy on HbA1c of 100 mg vildagliptin once daily as compared to placebo as add-on to metformin in patients with type 2 diabetes inadequately controlled with metformin.

ELIGIBILITY:
Inclusion Criteria:

* Patients on metformin for at least three months and on a stable dose of at least 1500 mg daily for a minimum of 4 weeks prior to visit 1
* Body mass index in the range 22-40
* Blood glucose criteria must be met

Exclusion Criteria:

* Pregnancy or lactation
* History of type 1 diabetes
* Evidence of significant diabetic complications

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2006-05; Primary Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c at 24 weeks | 24 weeks

SECONDARY OUTCOMES:
Safety of vildagliptin in combination with metformin during 24 weeks of treatment | 24 weeks
Change from baseline in fasting plasma glucose at 24 weeks | 24 weeks
Patients with endpoint HbA1c < 7% after 24 weeks | 24 weeks
Patients with reduction in HbA1c greater than or equal to 0.7% after 24 weeks | 24 weeks
Change from baseline in body weight at 24 weeks | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States
- Novartis Investigative Site, Investigative Centers, Germany

REFERENCES:
- [Result] Goodman M, Thurston H, Penman J. Efficacy and tolerability of vildagliptin in patients with type 2 diabetes inadequately controlled with metformin monotherapy. Horm Metab Res. 2009 May;41(5):368-73. doi: 10.1055/s-0028-1104604. Epub 2009 Feb 16. PMID 19221978